CLINICAL TRIAL: NCT05772988
Title: Examining the Effects of 3-weeks Beta-Alanine Supplementation on CrossFit® Performance
Brief Title: Beta-alanine Supplementation and CrossFit Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022_23_02
Record Dates: First submitted 2023-03-04; First posted 2023-03-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Exercise-Induced Lactic Acidemia
MeSH Terms: interventions — beta-Alanine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine (Experimental): Beta-alanine to be given for three weeks
  Interventions: Dietary Supplement: Beta-alanine
- Maltodextrin (Placebo Comparator): Placebo to be given for three weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Beta-alanine — Beta-alanine
  Arms: Beta-alanine
Dietary Supplement: Maltodextrin — Maltodextrin
  Arms: Maltodextrin

SUMMARY:
This study will randomize CrossFit participants to receive beta-alanine or placebo supplementation for 3 weeks. The study will be double-blind. Performance on the "Fran" test will be completed at baseline and after the 3 week intervention. Respiratory exchange ratio will also be assessed during the performance test at baseline and after 3 weeks.

DETAILED DESCRIPTION:
Beta-alanine is a nutritional supplement often consumed by people involved in high-intensity sports that involve substantial lactic acidosis. If consumed on a regular basis, it improves muscle buffering capacity and exercise performance during high-intensity moderate-duration events. CrossFit involves competitions that are high in intensity and moderate duration and many elite CrossFit athletes have reported taking beta-alanine as a supplement. It has never however been evaluated in a research study for its affect on CrossFit performance. The purpose of the study is therefore to assess the effects of beta-alanine supplementation on CrossFit performance. A maximum of 30 CrossFit participants will participate in this randomized double-blind parallel groups study. Participants will be randomized to receive 6.4 g/d beta-alanine or maltodextrin placebo for 3 weeks. At baseline and after the intervention, participants will complete a "Fran" test, which involves performing sets of repeated dumbbell thrusters alternating with chin-ups. The performance measure is the time to complete the test. During the test, respiratory exchange ratio will be assessed to indirectly assess acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of one year of CrossFit experience and doing CrossFit training at least twice a week

Exclusion Criteria:

* Having consumed beta-alanine in the past six months
* Having changed the dose of any other nutritional supplement within the past month
* Having suffered a major physical injury in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in time to perform a "Fran" CrossFit workout | Baseline, 3 weeks
  This involves alternating sets of dumbbell thrusters and pull-uips

SECONDARY OUTCOMES:
Change from baseline in respiratory exchange ratio | Baseline, 3 weeks
  Respiratory exchange ratio (carbon dioxide exhaled relative to oxygen consumed) during the performance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No